CLINICAL TRIAL: NCT06630754
Title: An Exploration of Body Composition in Older Adults Undergoing Systemic Anticancer Treatment.
Brief Title: Body Composition in Older Adults
Acronym: BODI
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CCR6064
Record Dates: First submitted 2024-09-19; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia in Elderly; Cachexia; Cancer; Sarcopenia; Body Composition Changes; Older Adults; Nutrition
MeSH Terms: conditions — Cachexia; Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adults aged 70yrs and older, eligible, and accepting of assessment in the SAOP.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention; observation cohort study

SUMMARY:
The primary aim of the study is to explore body composition in older adults (aged 70 years and over) with cancer, undergoing systemic anticancer treatment. Additional aims include to explore the extent of body composition changes and whether changes are tumour specific, the incidence for cancer-related cachexia and sarcopenia and finally, how body composition can inform nutritional management of older adults with cancer.

To do this, the investigators applied for and were awarded funding from a company called Nutricia to pay for a band 4 (0.6 WTE for 7 months) to take monthly body composition measures on the patients who are eligible, accepting of assessment by the Senior Adult Oncology Programme (SAOP) and consent to these measures. Measurements will include an analysis from the Bioelectrical Impedance Analysis (BIA) machine which will quantify fat, lean muscle, and water content; waist to hip ratio; handgrip strength; calf circumferences. Socio-demographic data will also be collected.

Descriptive data analysis will take place to explore possible trends and associations which may inform future research and drive even further personalised care for this growing and typically underrepresented in research, population.

ELIGIBILITY:
Inclusion Criteria:

* Adults eligible and accepting of assessment in the SAOP.

  1. adults aged 70 years and over
  2. a cancer diagnosis
  3. just starting SACT
  4. able to provide at least 2 data sets during the study period (baseline + at least 1 research clinic visit)
  5. willing and able to provide written informed consent

Exclusion Criteria:

* No further exclusions

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: adults aged 70 years and older, with a cancer diagnosis who are to receive systemic anti-cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Explore body composition in older adults with cancer starting SACT. | 7 months
  means and standard deviations (or medians and interquartile ranges if not normally distributed) of body composition measures taken from all participants at baseline/ first Research Clinic, analysed at end of study will quantify this objective.

SECONDARY OUTCOMES:
Explore the extent of body composition changes in older adults with cancer during SACT. | 7 months
  percentage change between body composition measures taken from all participants at baseline and during monthly Research Clinics, analysed at end of study will quantify this objective.

OTHER OUTCOMES:
Explore whether there are differences between body composition in older adults with cancer receiving SACT, based on tumour diagnosis | 7 months
  Tumour types will be categorised with frequencies reported. Means calculated from Exploratory Endpoint #2 of each category will be compared at end of study and quantify this objective.
Explore how body composition can inform nutritional management of older adults with cancer receiving SACT. | 7 months
  nutritional interventions provided (if any) will be categorised and cross-examined for correlations with mean percentage change in body composition (Outcome #2) at end of study to quantify this objective.
Investigate the incidence for cancer-related cachexia and sarcopenia in older adults with cancer receiving SACT. | 7 months
  standardised cut off values (World Health Organization, 2011; Cruz-Jentoft et al., 2019; Roeland et al., 2020) for indicating the presence of cancer-related cachexia and sarcopenia will be extracted from body composition measures taken from all participants at baseline and during monthly Research Clinics and presented as an overall frequency (of participants) and frequencies within each tumour type. Analysis will occur at end of study and will quantify this objective.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Eldridge, M.Sc. (Hons) Cancer Care Award, Study Director — Royal Marsden NHS Foundation Trust; Megan Pattwell, PGDip Dietetics, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, London, United Kingdom